CLINICAL TRIAL: NCT04170075
Title: A Novel Therapeutic Intervention to Restore Health and Functioning in Persons With Chemotherapy-Induced Peripheral Neuropathy
Brief Title: Whole Body Vibration for the Improvement of Health and Functioning in Participants With Chemotherapy-Induced Peripheral Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Kerri Winters, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00018342; NCI-2019-08961 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00018342 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2019-09-09; First posted 2019-11-20 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Chemotherapy-Induced Peripheral Neuropathy; Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (UC) (No Intervention): Participants randomly assigned to the UC group will serve as controls and will be tested at the same time points as the WBV group. The UC group will be asked not to change their physical activity or dietary habits across the intervention period and we will track any changes using a questionnaire.
- Whole body vibration (WBV) (Experimental): Participants assigned to the WBV group will participate in twice daily 10-minute WBV training sessions, 7 days a week. Each WBV session will consist of a series of timed stands on the vibration platform (Marodyne LiV). During a timed stand, participants will perform slow controlled weight shifting exercises and gentle squats. The vibration frequency will be set at 30Hz and the amplitude set at 50-200 microns, for a total body acceleration of 0.4g+/-20%.
  Interventions: Behavioral: Whole Body Vibration

INTERVENTIONS:
Behavioral: Whole Body Vibration — Undergo WBV
  Other Names: WBV; Whole Body Vibration Therapy
  Arms: Whole body vibration (WBV)

SUMMARY:
This clinical trial studies how well whole body vibration works in improving the health and functioning of participants with chemotherapy-induced peripheral neuropathy. Peripheral neuropathy is a condition caused by exposure to chemotherapy drugs that may involve numbness/tingling and/or pain in the hands and feet, which can have adverse effects on daily life. Whole body vibration may cause weight loss and improve mobility and pain levels in cancer survivors who report symptoms of peripheral neuropathy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the feasibility and safety of whole body vibration (WBV) in adult cancer survivors with chemotherapy-induced peripheral neuropathy (CIPN).

II. Determine the effect of WBV training on physical functioning in adult cancer survivors with CIPN.

III. Explore the effect of WBV training on symptom relief (neuropathy symptoms, pain, fatigue) and readiness to exercise in adult cancer survivors with CIPN.

OUTLINE: Participants are randomized to 1 of 2 groups.

GROUP I (WBV): Participants complete two 10-minute WBV sessions per day, 7 days per week for 12 weeks.

GROUP II (USUAL CARE [UC]): Participants receive usual care and keep their same physical activity or dietary habits over 12 weeks.

After completion of study treatment, participants are followed up at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed cancer stage I-IIIc (confirmed by self-report on the Health History Questionnaire. If the patient is unable to confirm, we will send a letter to their physician to confirm for this criterion)
* Previous chemotherapy within five years of enrollment (confirmed by self-report on the Health History Questionnaire. If the patient is unable to confirm, we will send a letter to their physician to confirm for this criterion)
* Presence of mild-very severe CIPN symptoms (confirmed by assessment using the Patient-Reported Outcomes [PRO]-Common Terminology Criteria for Adverse Events [CTCAE] criteria)
* Age 18 years or older at enrollment (confirmed by self-report on the Health History Questionnaire)

Exclusion Criteria:

* Body weight > 275 pounds (confirmed by self-report on the Health History Questionnaire)
* A medical condition, movement or neurological disorder, or medication use that contraindicates participation in low intensity exercise and/or WBV (confirmed by self-report on the Health History Questionnaire, and by physician clearance, if in the professional opinion of the Principal Investigator, Dr. Kerri Winters-Stone, contraindications other than those identified by the patient or physician are present, she may consider the participant ineligible.)
* Presence of any known metastases (confirmed by self-report on the Health History Questionnaire. If the patient is unable to confirm, we will send a letter to their physician to confirm for this criterion)
* Adjuvant treatment for cancer within previous six weeks, other than hormone blocking, targeted or immunotherapy (confirmed by self-report on the Health History Questionnaire. If the patient is unable to confirm, we will send a letter to their physician to confirm for this criterion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2022-12-09 (Actual)

PRIMARY OUTCOMES:
Accrual | Up to 12-weeks
  The number of participants enrolled during the recruitment period.
Adherence | Up to 12-weeks
  Adherence = % of sessions attended and compliance = % of each session completed.
Compliance | Up to 12-weeks
  Compliance = % of each session completed.
Adverse events | Weekly up to 12-weeks
  An in-house survey will ask about adverse events (e.g., bone pain, nausea) that occur during the intervention. The number of discrete moderate and severe adverse events will be summed as a single variable.

SECONDARY OUTCOMES:
Objective physical function | 0, 12 weeks
  Measured by the Physical Performance Battery (PPB) to determine a person's ability to perform daily tasks independently. The PPB consists of 3 timed tests: 5 repeated chair stands, standing balance, and gait speed over 4 meters. Each test is scored 0 (unable) to 4 (completes without difficulty), based on quartiles of performance, then scores are summed. The possible range of scores is 0-12.
Functional mobility | 0, 12 weeks
  Functional mobility will be measured by the Timed Up and Go (TUG) test which measures the time that it takes a person to rise from a chair, walk 7 m, turn around and return and sit in the chair.
Functional balance-sway velocity | 0, 12 weeks
  Functional balance will be measured by postural sway which evaluates how well a person can maintain their equilibrium during quiet standing. Will conduct a standard 30-second postural sway test to measure the sway velocity (m/s) during quiet standing with feet together and eyes closed using lightweight, inertial wireless sensors worn on the trunk.
Functional balance-sway area | 0, 12 weeks
  Functional balance will be measured by postural sway which evaluates how well a person can maintain their equilibrium during quiet standing. Will conduct a standard 30-second postural sway test to measure the sway area (m2/s3) of sway during quiet standing with feet together and eyes closed using lightweight, inertial wireless sensors worn on the trunk.
Functional balance-sway amount | 0, 12 weeks
  Functional balance will be measured by postural sway which evaluates how well a person can maintain their equilibrium during quiet standing. Will conduct a standard 30-second postural sway test to measure the amount (m/s2) of sway during quiet standing with feet together and eyes closed using lightweight, inertial wireless sensors worn on the trunk.
Symptoms of chemotherapy-induced peripheral neuropathy | 0, 12 weeks
  Chronic changes in symptoms will be assessed at 0 and 12 weeks using the Functional Assessment of Cancer Therapy Gynecologic Oncology Group Neurotoxicity (FACT/GOG-Ntx). The questionnaire consists of the 27 item FACT-G, plus 11 items that specifically measure chemotherapy-induced neuropathy symptoms and concerns. Higher scores indicate worse symptoms.
Fatigue Visual Analog Scale | Before and after every whole body vibration session, up to 2 times per day, 7 days per week, for 12 weeks
  Fatigue overall will be measured both before and after each whole body vibration session using a visual analog scale to identify any acute symptom relief from training. The scale ranges from 0 (no fatigue) to 10 (worst fatigue).
Patient Reported Outcomes Measurement Information System (PROMIS) fatigue scale | 0, 12 weeks
  Chronic changes in fatigue will be assessed using the PROMIS Fatigue Scale. This instrument includes 8 items rated on a 5 point scale from "not at all" to "very much". Higher scores indicate worse fatigue.
Pain Visual Analog Scale | Before and after every whole body vibration session, up to 2 times per day, 7 days per week, for 12 weeks
  Pain in the feet will be assessed both before and after each session using a visual analog scale to identify any acute symptom relief from training. The scale ranges from 0 (no pain) to 10 (worst pain).
Brief Pain Inventory | 0, 12 weeks
  Chronic changes in pain will be assessed using the Brief Pain Inventory (BPI). The instrument has 2 subscales: pain severity and pain interference. Severity is determined by the average of 4 items rated from 0 (no pain) to 10 (pain as bad as you can imagine). Pain interference is determined by the average of 7 items rated from 0 (does not interfere) to 10 (completely interferes).
Body mass index | 0, 12 weeks
  Body mass index will be calculated as kg/m2.
Exercise readiness | 1, 12 weeks
  Exercise readiness will be assessed using the stage of change for exercise questionnaire. This is a categorical instrument with 5 options that indicate a person's readiness to engage in regular physical activity. Options that suggest engagement in more regular exercise are better.
Perceived physical function | 0, 12 weeks
  Perceived physical function will be measured by self-report using the Late-Life Function and Disability Instrument (LLFDI).
Gait | 0, 12 weeks
  The number of meters that participants can walk in 6-minutes will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Kerri Winters-Stone, PhD, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
What data in particular will be shared? All individual quantitative participant data collected during the trial, after deidentification.
  What other documents will be available? None
  With whom? Investigators who provide a methodologically sound proposal and complete a data sharing agreement that includes commitments to: (1) using the data only for research purposes and not to identify any individual participant, (2) securing the data using appropriate computer technology, and (3) destroying or returning the data after analyses are completed.
  For what types of analyses? To achieve aims in the approved proposal.
Time Frame: Beginning 3 months following publication. No end date.
Access Criteria: Proposals should be directed to wintersk@ohsu.edu. To gain access to data, data requestors will need to sign a data sharing agreement and be approved to receive the data by the OHSU IRB.

REFERENCES:
- [Derived] Ernst M, Wagner C, Oeser A, Messer S, Wender A, Cryns N, Brockelmann PJ, Holtkamp U, Baumann FT, Wiskemann J, Monsef I, Scherer RW, Mishra SI, Skoetz N. Resistance training for fatigue in people with cancer. Cochrane Database Syst Rev. 2024 Nov 28;11(11):CD015518. doi: 10.1002/14651858.CD015518. PMID 39606939